CLINICAL TRIAL: NCT02954367
Title: Effects of Meat Protein Administration on Body Composition, Strength, Immunological, Microbiota and Haematological Markers in Endurance Athletes
Brief Title: Meat and Whey Protein Supplementation in Endurance Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Europea de Madrid (Other)
Collaborators: University of Greenwich (Other)
Responsible Party: Principal Investigator, DIEGO MORENO PÉREZ, PhD, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BEEF-UEM-01
Record Dates: First submitted 2016-10-19; First posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Dietary Modification
MeSH Terms: interventions — Proteins; Red Meat; Carbohydrates; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PROTEIN (MEAT + WHEY) (Experimental): Post workout (training days) or breakfast (non training days) 20g of meat protein (10g meat + 10g whey) mixed with 200ml of orange juice and water
  Interventions: Dietary Supplement: PROTEIN
- CARBOHYDRATE (CHO) (Placebo Comparator): Post workout (training days) or breakfast (non training days) 20g of maltodextrin mixed with 200ml orange juice and water
  Interventions: Dietary Supplement: CARBOHYDRATE

INTERVENTIONS:
Dietary Supplement: PROTEIN — Immediately (<10 min) after completing each training session (resistance training) participants will consume a beverage containing 20g of meat protein (10g) plus whey (10g) mixed with 200 ml of orange juice and water. On non-training days supplement will be ingested before breakfast.
  Other Names: 100% BEEF
  Arms: PROTEIN (MEAT + WHEY)
Dietary Supplement: CARBOHYDRATE — Immediately (<10 min) after completing each training session (resistance training), participants will consume a beverage containing about 20g of maltodextrin mixed with 200 ml of orange juice and water. On non-training days supplement will be ingested before breakfast.
  Other Names: Maltodextrin
  Arms: CARBOHYDRATE (CHO)

SUMMARY:
The aim of this project is to investigate the potential benefits of combining a new protein meat hydrolysates extract with a regular endurance training programme on (a) body composition (b) performance (c) muscle structure (d) immunology and (e) microbiota (f) haematological markers in endurance athletes

DETAILED DESCRIPTION:
PROYECT DESIGN This investigation involves a 10-week randomised, balanced, double blind parallel group between-subjects design, aimed to analyse the effects of combining endurance exercise and a post exercise nutrition strategy (hydrolysates meat protein (MEAT) + whey protein (W) or a isocaloric only carbohydrate placebo) on training outcomes, immunity and haematological variables after regular training and feeding intervention.

Participants will be divided in two-treatment groups 1) Hydrolysed meat-protein + whey (PROT); and 2) non-protein iso-energetic placebo (CHO). Once considered eligible for the study, and after an initial familiarisation period plus baseline tests (endurance performance body composition and blood extractions) participants will be randomly assigned to one of the intervention groups: PROT and CHO. Each group will follow a 10-week periodised endurance training intervention combined with one of the two specific supplementation treatments (PROT or CHO). Measurements of performance (VO2peak, vetilatory threshold and time to exhaustion at maximal aerobic intensity), body composition (fat and fat free mass), microbiota and haematology will be determined before and after the 10-week intervention period.

Once informed consent and health history have been obtained, after the baseline assessment (t1), participants will be divided into two similar profile groups, matched by body mass, age, sex and maximal oxygen uptake (VO2peak): (1) PROT (2) CHO

INTERVENTION The intervention will comprise of a 10-week combined supplementation (MEAT + W and CHO) regular endurance-training programme.

Endurance training Participants will commit to follow a polarised triphasic endurance-training model. This model contains three intensity zones calculated as low intensity [< the first ventilatory threshold (VT1), ~ 70% HRmax]; moderate intensity [between VT1 and respiratory compensation point or ventilatory threshold 2 (VT2), >70 < 90% HRmax]; and high intensity [>VT2, 90% HRmax]. Participants will train 5 to 6 times per week with a total percentage distribution of 75 to 80% at low intensity; 10% at moderate intensity, and 15 to 10% at high intensity.

Cardiorespiratory test Participants will perform a maximal cardiorespiratory exercise test before the training period to determine peak oxygen uptake (VO2peak) and ventilatory thresholds. Percentage of HRmax and the 15 points (6 to 20) Borg Scale Rate of Perceive Exertion (RPE) will be used to appropriately select the load along the training intervention.

Supplementation protocol Training days: Immediately (<10 min) after completing each training session, participants will consume a beverage containing 20g of supplement (10g MEAT + 10g W) plus 200 ml of orange juice or only carbohydrate placebo (maltodextrine and orange juice).

Non-training days: before breakfast.

Supplements and placebo will be provided in powder form and should be mixed with 200ml of orange juice and water at the moment of consumption.

The supplements and placebo will look and taste identical.

Thus a total of one 20g doses will be administered on a daily base. Participants are required to ingest a total of 70 for the total of 10 weeks of the study intervention.

Supplements will be provided in 14 days intervals and distributed by a blinded researcher after participants return the empty bag of the supplement/placebo consumed during the previous 14 day period.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 45
* Vo2max >50ml/kg/min
* Regularly trained athletes,
* Minimum 3 years of experience in resistance training exercise,
* Volunteers,

Exclusion Criteria:

* any musculoskeletal injuries, metabolic conditions, or diseases;
* use of medications, smoking, and nutritional supplements known to affect physical performance, muscle damage or recovery process (e.g., creatine, whey protein, and amino acids) within 6 weeks prior to the start of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
% Fat Mass (Body composition) | 10 weeks
  Estimated with Densitometry (DEXA)
Visceral Adipose Tissue Mass (g) (Body composition) | 10 weeks
  Estimated with DEXA
Total Fat Free mass (g) (Body composition) | 10 weeks
  Estimated with DEXA
Bone mineral density (g/cm3) (Body composition) | 10 weeks
  Estimated with DEXA

SECONDARY OUTCOMES:
Blood Glucose (mg/dl) | 10 weeks
Creatine Kinase (Ul/l) -Blood markers- | 10 weeks
Creatinine (mg/dl) - Blood markers - | 10 weeks
Myoglobin (ng/ml) - Blood markers - | 10 weeks
Total cholesterol (mg/dl) -Blood markers- | 10 weeks
HDL cholesterol (mg/dl) -Blood markers- | 10 weeks
LDL cholesterol (mg/dl) -Blood markers- | 10 weeks
Aspartate amino transferasa (Ul/l) -Blood markers- | 10 weeks
Triglycerides (mg/dl) -Blood markers- | 10 weeks
Hemoglobin (g/dl) -Blood markers- | 10 weeks
Erythrocyte (M/µL) -Blood markers- | 10 weeks
Haematocrit (%) -Blood markers- | 10 weeks
Mean corpuscular volume (cubic millimeter)-Blood markers- | 10 weeks
Serum Transferrin (mg/dl) -Blood markers- | 10 weeks
Transferrin saturation (%) -Blood markers- | 10 weeks
Neutrophils (%) -Blood markers- | 10 weeks
Lymphocyte (%) -Blood markers- | 10 weeks
Monocytes (%) -Blood markers- | 10 weeks
Ferritin, serum (ng/ml) -Blood markers- | 10 weeks
Progressive maximal oxygen consumption test (Cardiorespiratory test) | 10 weeks
  - Maximum oxygen uptake (ml/kg/min)
Time to exhaustion at maximal aerobic (min) | 10 weeks
Gut microbiota determination by 16S rRNA Sequencing | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: DIEGO MORENO, PhD, Principal Investigator — Universidad Europea de Madrid; FERNANDO NACLERIO, PhD, Principal Investigator — University of Greenwich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moreno-Perez D, Lopez-Samanes A, Larrosa M, Larumbe-Zabala E, Centeno A, Roberts J, Naclerio F. Effects of protein-carbohydrate vs. carbohydrate alone supplementation on immune inflammation markers in endurance athletes: a randomized controlled trial. Eur J Appl Physiol. 2023 Jul;123(7):1495-1505. doi: 10.1007/s00421-023-05168-6. Epub 2023 Mar 14. PMID 36918416